CLINICAL TRIAL: NCT05996861
Title: Multidisciplinary Protocol for Best Pracrice in Sleep for Critically Ill Patients
Brief Title: Protocol For Sleep for Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Moinhos de Vento (Other)
Responsible Party: Principal Investigator, Laura Drehmer, Principal investigator, Hospital Moinhos de Vento
Other Study IDs: 842
Record Dates: First submitted 2023-07-10; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Sleep Disorders
Keywords: Sleep; ICU; Delirium; Multidisciplinary Team; Sleep Protocol
MeSH Terms: conditions — Sleep Wake Disorders; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-sleep protocol group: Patients with inclusion criteria assessed before the implementation of the sleep protocol.
- Post-sleep protocol group: Patients with inclusion criteria after the implementation of the sleep protocol.
  Interventions: Behavioral: ICU sleep protocol

INTERVENTIONS:
Behavioral: ICU sleep protocol — Adjusting sound intensity, as well as reducing noise: efforts will be made to minimize staff conversation volume during the night.
  Earplugs will be offered, along with the provision of eye masks for lucid patients, and thermal comfort adjustments will be made, such as providing blankets and/or adjusting room temperature.
  Dimming of lights starting from 10 PM. Reduced circulation of external services between 11 PM and 6 AM, and rationalization of sample collections and/or patient transfers between beds during the 11 PM to 6 AM interval.
  Optimization of analgesics for better pain control; optimization of medication use during wakefulness when clinically feasible; adjustment of intervals for capillary blood glucose measurement; maintaining and/or resuming the use of chronic sleep medications. If the patient has been unable to sleep, a hypnotic medication will be offered.
  Other considerations include suggesting ventilatory support measures for selected patients.
  Groups: Post-sleep protocol group

SUMMARY:
Sleep is essential for health and well-being. The quality of sleep impacts physical and cognitive aspects, including memory, immune system, and neuroendocrine function, with abnormalities associated with cardiovascular changes, neuropsychiatric disorders, and mortality. Additionally, sleep disorders are related to an increased incidence of delirium in Intensive Care Units (ICUs). Routines to control environmental factors in ICUs seem to have an impact on reducing the incidence of acute brain dysfunction - delirium - and could help prevent sleep disturbances in critically ill patients. This study aims to demonstrate an improvement in sleep quality in critically ill patients through the reduction of the Richards-Campbell Sleep Questionnaire score and propose a package of measures to improve sleep practices in ICU-admitted patients.

DETAILED DESCRIPTION:
Detailed description:

Critically ill patients are particularly vulnerable to sleep disorders. In the context of critical illness and ICU admission, there is an intersection of factors contributing to this situation: pre-existing health conditions, severe acute illness, sleep-altering treatments (sedatives, analgesics, mechanical ventilation), psychiatric disorders, and the physical environment. In addition to the impact during hospitalization, the literature points to a long-term reduction in quality of life due to sleep disturbance. Recent studies following up on patients after ICU discharge reveal high rates of sleep disorders up to 6 months after hospital discharge - related or unrelated to new psychiatric disorders and even cognitive changes. Furthermore, sleep disorders are associated with an increased incidence of delirium in ICUs, which refers to altered consciousness and cognition in patients admitted to the intensive care environment, which are associated with worsened patient outcomes such as increased hospital stay and consequently the risk of fatal complications. The prevalence of delirium is around 70%, with an incidence of 89%. Delirium assessment in ICUs is usually performed daily.

In order to improve the sleep quality of this population, there are modifiable factors, whether environmental (lighting, noise, general care), physiological (medications, ventilatory parameter adjustments), or psychological (anxiety, pain, absence of family members). Routines to control environmental factors in ICUs seem to have an impact on reducing the incidence of acute brain dysfunction - delirium - and could help prevent sleep disturbances in critically ill patients. These measures include dimming or reducing corridor lights at night, grouping (when possible) care activities at appropriate times, raising curtains, and encouraging mobilization during daytime shifts. For non-delirious patients, the use of earplugs and eye masks is also recommended.

Therefore, the investigators have developed this research project with the aim of evaluating the implementation of a multifaceted and multidisciplinary protocol to promote an improvement in sleep quality in critically ill patients.

The SPIRIT Protocol is a summary of recommendations for clinical trials, which was used as a support in this study. This is a multicenter clinical trial with a quasi-experimental design.

The first step consists of assessing the sleep quality in sequential patients admitted to the ICU and characterizing the disruptive elements.

After this period, the second step will involve sensitizing and training the multidisciplinary team about the importance of sleep for critically ill patients and providing training for the implementation of a multifaceted protocol of interventions to promote sleep quality improvement.

Once the multidisciplinary protocol is implemented, the sleep quality of the patients and the clinical impact of this protocol will be reevaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older);
* Have spent at least two nights in the ICU;
* Neuropsychiatric conditions to respond to the sleep questionnaire Informed consent - authorization through the ICF (Informed Consent Form).

Exclusion Criteria:

* Neuropsychiatric conditions that prevent responding to the questionnaire, such as patients with dementia, severe sequelae of cerebrovascular disease, inability to understand and/or communicate, severe encephalopathy, deep sedation, acute brain dysfunction and/or delirium, visual and/or auditory acuity impairments that prevent responding to the questionnaire, active alcoholism, active illicit drug use, severe withdrawal symptoms;
* Patients with deep sedation that does not allow interaction with the evaluator;
* Moribund patients;
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the intensive care unit with a minimum stay of two nights
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Richards-Campbell Sleep Quality Score | before and one month after implementation of the sleep protocol
  To demonstrate a better sleep quality in critical patients

SECONDARY OUTCOMES:
Change in the Sleep in the ICU Questionnaire | before and one month after implementation of the sleep protocol
  Characterization of the perception of factors influencing sleep in critically ill patients
Change in the Confusion Assessment Method for the ICU | before and one month after implementation of the sleep protocol
  To evaluate the incidence of delirium and its duration according to sleep quality;
Change in the Questionnaire on the patient's perception of sleep from the family member's point of view | before and one month after implementation of the sleep protocol
  To compare patient satisfaction at ICU discharge with family satisfaction
Change in the Questionnaire for the evaluation of the multidisciplinary team regarding prior knowledge of sleep protocol | before implementation of the sleep protocol
  To assess the knowledge of the multidisciplinary team regarding sleep in critically ill patients before the implementation of the multidisciplinary protocol
Change in the Questionnaire for assessing and perceiving patients' sleep from the point of view of the care team | one month after implementation of the sleep protocol
  To assess the perception of the multidisciplinary team regarding the sleep quality of hospitalized patients after the implementation of the multidisciplinary protocol
Change in the Pittsburgh Sleep Quality Index and Epworth Sleepiness Scale. | at three and six months after hospital discharge
  To evaluate the sleep quality of surviving patients of critical illnesses at ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Laura Drehmer, Principal Investigator — Vale dos Sinos Hospital; Felippe Dexheimer, Study Director — Moinhos de Vento Hospital; Cassiano Teixeira, Study Director — Moinhos de Vento Hospital
Locations (2):
- Brazil (2):
  - Unimed Vale dos Sinos Hospital, Novo Hamburgo, Rio Grande do Sul
  - Moinhos de Vento Hospital, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altman MT, Knauert MP, Pisani MA. Sleep Disturbance after Hospitalization and Critical Illness: A Systematic Review. Ann Am Thorac Soc. 2017 Sep;14(9):1457-1468. doi: 10.1513/AnnalsATS.201702-148SR. PMID 28644698
- [Background] Beltrami FG, John AB, de Macedo BR, Correa Junior V, Nguyen XL, Pichereau C, Maury E, Fleury B, Gus M, Fagondes SC. A multi-intervention protocol to improve sleep quality in a coronary care unit. Eur J Cardiovasc Nurs. 2022 Jun 30;21(5):464-472. doi: 10.1093/eurjcn/zvab099. PMID 34935040
- [Background] Ritmala-Castren M, Virtanen I, Vahlberg T, Leivo S, Kaukonen KM, Leino-Kilpi H. Evaluation of patients' sleep by nurses in an ICU. J Clin Nurs. 2016 Jun;25(11-12):1606-13. doi: 10.1111/jocn.13148. Epub 2016 Mar 18. PMID 26991592
- [Background] Ebben MR, Spielman AJ. Non-pharmacological treatments for insomnia. J Behav Med. 2009 Jun;32(3):244-54. doi: 10.1007/s10865-008-9198-8. Epub 2009 Jan 24. PMID 19169804
- [Background] Mori S, Takeda JR, Carrara FS, Cohrs CR, Zanei SS, Whitaker IY. Incidence and factors related to delirium in an intensive care unit. Rev Esc Enferm USP. 2016 Jul-Aug;50(4):587-593. doi: 10.1590/S0080-623420160000500007. English, Portuguese. PMID 27680043
- [Background] Richards KC, Wang YY, Jun J, Ye L. A Systematic Review of Sleep Measurement in Critically Ill Patients. Front Neurol. 2020 Nov 6;11:542529. doi: 10.3389/fneur.2020.542529. eCollection 2020. PMID 33240191
- [Background] Telias I, Wilcox ME. Sleep and Circadian Rhythm in Critical Illness. Crit Care. 2019 Mar 9;23(1):82. doi: 10.1186/s13054-019-2366-0. PMID 30850003
- [Result] Li SY, Wang TJ, Vivienne Wu SF, Liang SY, Tung HH. Efficacy of controlling night-time noise and activities to improve patients' sleep quality in a surgical intensive care unit. J Clin Nurs. 2011 Feb;20(3-4):396-407. doi: 10.1111/j.1365-2702.2010.03507.x. PMID 21219521
- See also: SPIRIT 2013 Checklist — http://www.spirit-statement.org/spirit-statement/

DOCUMENTS (2):
  • Statistical Analysis Plan (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT05996861/SAP_000.pdf
  • Informed Consent Form (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT05996861/ICF_001.pdf